CLINICAL TRIAL: NCT03443804
Title: A Multicenter, Randomized, Double-blinded, Parallel, Active-controlled, Phase 3 Clinical Trial to Evaluated the Efficacy and Safety of DW-1401 in Acute and Chronic Gastritis Patients
Brief Title: To Evaluate the Efficacy and Safety of DW-1401 in Acute and Chronic Gastritis Patients
Acronym: 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DW1401-302
Record Dates: First submitted 2018-02-11; First posted 2018-02-23 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Gastritis Acute; Gastritis Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test(DW1401) (Experimental): tid PO, DW1401+Placebo of Stillen tab.
  Interventions: Drug: Test(DW1401)
- Reference(Stillen tab.) (Active Comparator): tid PO, Stillen tab.+Placebo of DW1401
  Interventions: Drug: Reference(Stillen tab.)

INTERVENTIONS:
Drug: Test(DW1401) — DW1401+Placebo of Stillen tab.
  Arms: Test(DW1401)
Drug: Reference(Stillen tab.) — Stillen tab.+Placebo of DW1401
  Arms: Reference(Stillen tab.)

SUMMARY:
Evaluate the Efficacy and Safety of DW1401 versus Stillen tab. in Patients with Acute or Chronic Gastritis

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with acute or chronic gastritis in a gastroscopy performed within 7 days prior to administration of this trial.
* At least one or more erosions have been identified on gastroscopy.
* Patients who decided to voluntarily participate in this trial and agreed in writing.

Exclusion Criteria:

* Patients who can not undergo gastroscopy
* Peptic ulcer (except scarring) and reflux esophagitis
* Patients who have had gastric acid suppression surgery or stomach/esophagus surgery (except for simple perforation surgery and appendectomy)
* Patients with a history of gastrointestinal malignancies
* Zollinger-Ellison syndrome patients
* Patient with spontaneous coagulation disorder
* Patients with an allergic or hypersensitive response to a study drug
* Patients with a potential pregnancy.
* Patients who had clinically significant abnormalities in the screening test. (ALT, AST, BUN, Serum creatinine is more than twice the upper limit)
* Pregnant and lactating women
* Those currently taking other study drugs
* patients who were judged to be ineligible for the trial by the principle investigator and the person in charge.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The efficacy rate on gastroscopy | 0, week 2
  The efficacy rate is obtained from the following formula using the subject whose erroneous score is improved by 50% or more as compared with before the study drug administration.
  The efficacy rate(%) = (number of effective cases)/(all cases) x 100
  Effective case is determined by the grade change of erosion. A case in which the grade changes from 4 to 2 or 1, from 3 to 1, or from 2 to 1 is judged as an effective case.

SECONDARY OUTCOMES:
Cure rate on gastroscopy | 0, week 2
  Judging from the gastroscopic examination as normal (no erosion), the cure rate is obtained as follows.
  Cure rate(%) = (number of cures(no erosion))/(all cases) x 100

IPD SHARING:
Plan to Share IPD: No
There is no plan for IPD.